CLINICAL TRIAL: NCT00920881
Title: Protocol #TS05-066 Clinical Evaluation of the Accuracy of the FreeStyle Navigator Continuous Glucose Monitoring System
Brief Title: Clinical Evaluation of the Accuracy of the FreeStyle Navigator Continuous Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Deryck Wade, Director Clinical Affairs, Abbott Diabetes Care
Other Study IDs: TS05-066
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus
Keywords: Continuous glucose monitoring; Accuracy; Continuous glucose-error grid analysis
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes
  Interventions: Device: FreeStyle Navigator Continuous Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Navigator Continuous Glucose Monitoring System — Subjects wore 2 Navigator sensors for approximately 122 hours. Subjects and clinical staff were masked to continuous glucose data. During the time the subjects wore the continuous sensor, they were instructed to continue with their current diabetes management plan. Subjects stayed at the clinic for approximately 50 hours during the study period. While in the clinic, venous blood samples were collected every 15 minutes to determine whole blood reference glucose concentrations using the Yellow Springs Instrument. Subjects were also asked to obtain up to 50 FreeStyle finger blood glucose measurements using the system in the Navigator receiver for comparative analysis and system calibration. This was not a treatment study.

SUMMARY:
To evaluate the clinical accuracy of the FreeStyle Navigator Continuous Glucose Monitoring System with respect to a reference standard.

ELIGIBILITY:
Inclusion Criteria:

* History consistent with type 1 diabetes
* At least 18 years of age
* Available and capable of following the protocol instructions provided by the healthcare professional
* Signed and dated informed consent form

Exclusion Criteria:

* Pregnancy
* Type 2, gestational, or secondary diabetes
* Known allergy to medical grade adhesives
* Skin abnormalities at the insertion sites that would confound the assessment of the effect of the device on the skin
* Seizure disorder
* Myocardial ischemia
* History of stroke
* Severe hypoglycemia unawareness
* Other concomitant medical conditions that in the opinion of the investigator, would affect the evaluation of device performance and/or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects recruited from clinical research centers which specialize in diabetes-related therapies.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Bugler, Study Director — Abbott Diabetes Care
Locations (3):
- United States (3):
  - Diablo Clinical Research, Walnut Creek, California
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas
  - Ranier Clinical Research, Renton, Washington

REFERENCES:
- [Result] Weinstein RL, Schwartz SL, Brazg RL, Bugler JR, Peyser TA, McGarraugh GV. Accuracy of the 5-day FreeStyle Navigator Continuous Glucose Monitoring System: comparison with frequent laboratory reference measurements. Diabetes Care. 2007 May;30(5):1125-30. doi: 10.2337/dc06-1602. Epub 2007 Mar 2. PMID 17337488
- [Result] McGarraugh G, Bergenstal R. Detection of hypoglycemia with continuous interstitial and traditional blood glucose monitoring using the FreeStyle Navigator Continuous Glucose Monitoring System. Diabetes Technol Ther. 2009 Mar;11(3):145-50. doi: 10.1089/dia.2008.0047. PMID 19216686